CLINICAL TRIAL: NCT01175265
Title: Effects of Breathing Retraining on Pulmonary Function, Exercise Capacity, Quality of Life and Cardiac Autonomic Function in Patients With COPD
Brief Title: Effects of Breathing Retraining in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Prof. Dr. dipl. Ing. H. Teschler, Ruhrlandklinik
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDAAA
Record Dates: First submitted 2010-07-13; First posted 2010-08-04 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: clinically stable; COPD (GOLD-classification I-IV); COPD; breathing retraining; pulmonary rehabilitation; cardiac autonomic function; quality of life; exercise capacity; pulmonary function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pulmonary rehabilitation, no breathing retraining (No Intervention): Forty COPD patients (23 females) with a mean (SD) age of 66.0 (6.3) years and a FEV1 of 47.1 (18.9) % predicted were randomized to conventional pulmonary rehabilitation (n=20) and conventional pulmonary rehabilitation plus breathing retraining (n=20).
- breathing retraining (No Intervention): Forty COPD patients (23 females) with a mean (SD) age of 66.0 (6.3) years and a FEV1 of 47.1 (18.9) % predicted were randomized to conventional pulmonary rehabilitation (n=20) and conventional pulmonary rehabilitation plus breathing retraining (n=20).
  Interventions: Other: respiratory biofeedback

INTERVENTIONS:
Other: respiratory biofeedback — In order to train effortless diaphragmatic breathing techniques the biofeedback loop starts at the sensor that measures the patient's breathing rhythm at both umbilical and abdominal level. The sensor is connected to an amplifier that converts the electrical impulses into acoustical and visual outputs. Patients were encouraged to regulate their breathing patterns at a 10-20% slower respiration rate resulting in increased tidal volumes. Furthermore, the patients were encouraged to reduce dynamic hyperinflation by completing the expiration prior to the initiation of the next breath while using pursed-lips breathing. Patients were trained to breath as comfortable as possible with predominant abdominal expansion during the inhalation and smooth abdominal contraction during exhalation.
  Arms: breathing retraining

SUMMARY:
Conventional pulmonary rehabilitation programs improve exercise tolerance, peripheral muscle strength, and health related quality of live but not pulmonary function in patients with chronic obstructive pulmonary disease (COPD). The role of breathing retraining techniques in the rehabilitation of patients with COPD remains unclear. The hypothesis to be tested in this study is that pulmonary function, cardio-pulmonary exercise capacity, health related quality of life and cardiac autonomic modulation of patients with COPD who undergo pulmonary rehabilitation plus breathing retraining will be better than that of patients undergoing a conventional pulmonary rehabilitation.

DETAILED DESCRIPTION:
To address this uncertainty, we performed a randomized controlled trial to assess the effects of a 4-week rehabilitation program including breathing retraining on pulmonary function (PFT), cardio-pulmonary exercise capacity (CPET), health related quality of life (HRQL) and cardiac autonomic modulation (CAM).

A randomized controlled trial comparing the effects of a conventional 4-week pulmonary rehabilitation program with those of a 4-week pulmonary rehabilitation program plus breathing retraining on pulmonary function (FEV1), cardiopulmonary exercise capacity (6-minute walking distance, 6MWD), health related quality of life (chronic respiratory questionnaire, CRQ) and cardiac autonomic function (rMSSD) was performed.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable patients with COPD (GOLD-classification I-IV)

Exclusion Criteria:

* Patients with clinical signs of COPD exacerbation
* Cardiac arrhythmia
* Coronary artery disease
* Primary pulmonary vascular disease
* Oxygen desaturation to less than 80% during exercise on room air

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
cardiopulmonary exercise capacity
  6-minute walking distance, 6MWD

SECONDARY OUTCOMES:
pulmonary function
  pulmonary function (FEV1)
quality of life
  health related quality of life (chronic respiratory questionnaire, CRQ)
autonomic function
  cardiac autonomic function (rMSSD)

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Teschler, Prof. Dr. dipl Ing, Study Director — Ruhlrandklink Essen
Locations (1):
- University Hospital Ruhrlandklinik, Essen, Nordrheinwestfalen, Germany

REFERENCES:
- [Derived] van Gestel AJ, Kohler M, Steier J, Teschler S, Russi EW, Teschler H. The effects of controlled breathing during pulmonary rehabilitation in patients with COPD. Respiration. 2012;83(2):115-24. doi: 10.1159/000324449. Epub 2011 Apr 7. PMID 21474911